CLINICAL TRIAL: NCT00825786
Title: Ultrasound Guided Supraclavicular Nerve Block: Comparison Between a Mixture of Mepivacaine and Ropivacaine, and Sequential Injection of Mepivacaine Followed by Ropivacaine
Brief Title: Ultrasound Guided Supraclavicular Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-671
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Local Anesthetic
Keywords: surgery for arm hand or elbow; mepivacaine; ropivacaine; hand surgery; elbow surgery; forearm surgery
MeSH Terms: interventions — Ropivacaine; Mepivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): combined group: ropivacaine and mepivacaine mixture: 1:1 volume mixture of 1.5% mepivacaine and 0.5% ropivacaine in 2 syringes (labeled 1 and 2) with 15 mL in each (total, 30 mL) injected in immediate sequence;
  Interventions: Drug: Ropivacaine; Drug: Mepivacaine
- Group 2 (Active Comparator): sequential group: mepivacaine followed by ropivacaine: syringe 1 containing 15 mL of 1.5% mepivacaine, syringe 2 containing 15 mL of 0.5% ropivacaine (total, 30 mL); syringe 2 was injected with a 90-sec delay after injection of syringe 1.
  Interventions: Drug: Ropivacaine; Drug: Mepivacaine

INTERVENTIONS:
Drug: Ropivacaine — ropivacaine (15 ml).
Drug: Mepivacaine — One syringe will contain mepivacaine (15 ml)

SUMMARY:
This study will test the hypothesis that sequential injection of 1.5% mepivacaine followed 90 seconds later by 0.5% ropivacaine in ultrasound guided supraclavicular block provides a quicker onset and a longer duration of analgesia than an equi-dose mixture of the two local anesthetics.

DETAILED DESCRIPTION:
Patients will be randomized into one of two groups, Group M: Ropivacaine and Mepivacaine - subject will receive two injections before surgery begins. These two injections will consist of the mixture of mepivacaine (15 ml) and ropivacaine (15 ml).

Group S: Mepivacaine followed by Ropivacaine. Subjects will receive two injections before surgery begins. One injection will contain mepivacaine (15 ml) and the other will contain ropivacaine (15 ml).

On the first, second, and third mornings after surgery,subjects will be asked to rate their pain on a scale of 1 to 10. If the subject is discharged from the hospital, a telephone call will be made to the subject's home to collect this information.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper extremity procedures suitable for supraclavicular anesthesia, including but not limited to oHand surgery oForearm surgery oElbow surgery
* Age between 18 and 70 years

Exclusion Criteria:

* Contraindications to supraclavicular block

  * Coagulopathy
  * Infection at the needle insertion site
  * Severe chronic obstructive pulmonary disease (COPD)
  * Contralateral pneumothorax or diaphragmatic paralysis
* Pregnancy
* Preexisting neuropathy involving the surgical limb
* Routine opioid use
* Inability to attain adequate ultrasound images in the supraclavicular area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Ritchey, MD, Principal Investigator — Cleveland Clinid; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: combined group: ropivacaine and mepivacaine mixture: 1:1 volume mixture of 1.5% mepivacaine and 0.5% ropivacaine in 2 syringes (labeled 1 and 2) with 15 mL in each (total, 30 mL) injected in immediate sequence;
  Ropivacaine: ropivacaine (15 ml).
  Mepivacaine: One syringe will contain mepivacaine (15 ml)
- Control: sequential group: mepivacaine followed by ropivacaine: syringe 1 containing 15 mL of 1.5% mepivacaine, syringe 2 containing 15 mL of 0.5% ropivacaine (total, 30 mL); syringe 2 was injected with a 90-sec delay after injection of syringe 1.
  Ropivacaine: ropivacaine (15 ml).
  Mepivacaine: One syringe will contain mepivacaine (15 ml)
Period: Overall Study
Arm/Group | Treatment | Control
Started | 52 | 51
Completed | 52 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13) | 46 (14) | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 27 | 19 | 46

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia.
Description: The primary outcomes will be the onset time, onset of surgical block, and duration of analgesia.
Time Frame: During surgery: postoperative day 0
Measure: Median (Inter-Quartile Range); unit: minute
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
minute | 7.5 [4 to 14] | 10 [7 to 20]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.14, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.46 to 1.09] — group 2 vs. group 1 (sequential vs combined)

2. Secondary Outcome: Time to Complete Motor Block
Time Frame: during surgery from induction time to end case time
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
minutes | 10 [5 to 18] | 19 [8 to 29]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.02, Log Rank

3. Secondary Outcome: Time to Onset of First Sensory Block
Time Frame: during surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
minutes | 0 [0 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.66, Log Rank

4. Secondary Outcome: Maximum Verbal Response Score (VRS) With Rest
Description: The severity of postoperative pain was assessed by an observer blinded to treatment using a 0- to 10-point verbal response score (VRS): 0 = no pain and 10= worst pain
Time Frame: through post operative day 3
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
mm | 4 [2 to 7] | 4 [1 to 6]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.60, ANCOVA

5. Secondary Outcome: Maximum Verbal Response Score (VRS) With Movement
Description: The severity of postoperative pain was assessed by an observer blinded to treatment using a 0- to 10-point verbal response score (VRS): 0 = no pain and 10 = worst
Time Frame: through post operative day 3
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
mm | 5.5 [3.5 to 8] | 5 [2 to 7]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.34, ANCOVA

6. Secondary Outcome: Duration of Analgesia
Description: Time from the complete onset of sensory block until first request for an analgesic
Time Frame: from surgery date to postoperative day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
hours | 9 [6 to 22] | 11 [7 to 20]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.15, Log Rank

7. Secondary Outcome: Total Opioid Consumption
Description: In morphine equivalent dose
Time Frame: postoperative day 1 to day 3
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 51
mg | 38 [11 to 90] | 30 [8 to 83]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.88, ANCOVA

ADVERSE EVENTS:
Time Frame: after surgery to hospital discharge
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No